CLINICAL TRIAL: NCT04188301
Title: Safety and Efficacy of Combination Therapy With Ivermectin, Diethylcarbamazine, and Albendazole (IDA) for Individuals With Onchocerciasis
Brief Title: Safety and Efficacy of IDA for Onchocerciasis
Acronym: DOLF IDA/Oncho
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Case Western Reserve University (Other); University of Health and Allied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201910085
Record Dates: First submitted 2019-12-02; First posted 2019-12-05 (Actual); Results first posted 2023-05-10 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Onchocerciasis
Keywords: ophthalmology
MeSH Terms: conditions — Onchocerciasis | interventions — Albumins

STUDY DESIGN:
Intervention Model Description: Participants will be split into two strata - those without ocular Mf detected six months after ivermectin pretreatment in the Part I preceding study AND without ocular Mf detected at baseline in the part II study will be in stratum 1. Those participants with ocular Mf detected 6 months after ivermectin pretreatment in the preceding study OR with ocular Mf detected at the baseline exam for this study will be in stratum 2. Stratum 1 will be enrolled first, followed by stratum 2. Members of each stratum will be evenly randomized into one of three treatment arms:
  1. IVM + ALB - Single dose of oral IVM (150 µg/kg) plus ALB (400 mg) (IVM/ALB)
  2. IDA x 1 dose - Single dose of oral IVM (150 µg/kg), DEC (6 mg/kg) and ALB (400 mg)
  3. IDA x 3 doses -Once daily for 3 days oral IVM (150 µg/kg), DEC (6 mg/kg) and ALB (400 mg)
Masking Description: While this is an open label study and there is no placebo treatment group, all efforts will be made to ensure that that medical/technical staff assessing skin Mf, adverse events (AEs) and ophthalmological findings will be unaware of initial baseline skin and ocular Mf findings and treatment arm as best as possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- IVM + ALB (Active Comparator): Single dose of oral IVM (150 µg/kg) plus ALB (400 mg)
  Interventions: Drug: IVM w/ ALB
- IDA x 1 dose (Experimental): Single dose of oral IVM (150 µg/kg), DEC (6 mg/kg) and ALB (400 mg)
  Interventions: Drug: Single dose of IDA
- IDA x 3 doses (Experimental): Once daily for 3 days oral IVM (150 µg/kg), DEC (6 mg/kg) and ALB (400 mg)
  Interventions: Drug: Three daily doses of IDA

INTERVENTIONS:
Drug: IVM w/ ALB — Participants will be given a single dose of oral IVM (150 µg/kg) plus ALB (400 mg) (IVM/ALB)
  Other Names: IA
  Arms: IVM + ALB
Drug: Single dose of IDA — Participants will be given a single dose of oral IVM (150 µg/kg), DEC (6 mg/kg) and ALB (400 mg)
  Other Names: IVM/DEC/ALB (x1)
  Arms: IDA x 1 dose
Drug: Three daily doses of IDA — Participants will be given one daily dose for 3 days of oral IVM (150 µg/kg), DEC (6 mg/kg) and ALB (400 mg)
  Other Names: IVM/DEC/ALB (x3)
  Arms: IDA x 3 doses

SUMMARY:
This DOLF study will investigate the safety and effectiveness of IDA treatment in persons with onchocerciasis when it is administered after pre-treatment with ivermectin to clear or greatly reduce microfilariae from the skin and eyes.

DETAILED DESCRIPTION:
This study will provide preliminary data on the safety of IDA treatment in persons with onchocerciasis when it is administered after pre-treatment with IVM to clear or greatly reduce microfilariae from the skin and eyes. Widespread use of IDA following IVM pretreatment (I/IDA) has the potential to greatly accelerate elimination of lymphatic filariasis (LF) in African countries that are co-endemic for LF and onchocerciasis. study later.

This study will also assess the efficacy of IDA for killing and sterilizing adult filarial worms. An improved macrofilaricidal treatment would be a major advance for the global program to eliminate onchocerciasis. Since the safety and efficacy objectives are both very important, we have included dual primary objectives for the study.

Primary objectives:

* Safety: To compare rates and types of severe adverse events (grade 3 or higher) that occur within 7 days following 1 day or 3 days of treatment with triple drug treatment ("IDA" = diethylcarbamazine (DEC) with ivermectin (IVM) and albendazole (ALB)) with the comparator regimen of 1 day of treatment with ivermectin and albendazole (IA) in persons with active Onchocerca volvulus infections after pretreatment with ivermectin alone.
* Efficacy: To compare the effect of three treatment regimens (1 day of IDA, 3 days of IDA, or IA) for killing or sterilizing adult female O. volvulus worms based on the percentage of all adult female worms in nodules that are alive with embryos in the uterus 18 months after treatment.

This is an open label, randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who were previously enrolled in the preceding Part I study (Protocol ID#201804116) and residing in the study area
* Must have at least palpable subcutaneous nodule (onchocercoma)
* Participants with baseline skin Mf counts less than or equal to 3 Mf/mg at the time of enrollment into the Part I study (Protocol ID#201804116)

Exclusion Criteria:

* Pregnant and breastfeeding mothers within 1 month of giving birth
* Severe eye disease at baseline including uveitis, severe glaucoma, severe keratitis, and/or cataracts that interfere with visualization of the posterior segment of the eye as well as the list of ocular diseases as outlined below. All ocular disease exclusion criteria apply to either eye. Bilateral disease is not necessary to exclude a participant. A participant will be excluded if any of the criteria are met for one eye.

  1. Any cataract of any type preventing clear visualization of fundus or imaging on Optical Coherence Tomography (OCT).
  2. Severe retinal nerve fiber layer thinning in the superior and inferior quadrant analysis on Ocular Coherence Tomography of the optic nerve with a corresponding visual field defect of grade 2 or worse on the same eye.If Ocular Coherence Tomography is not available, the following exclusion criteria will apply: vertical Cup/disc ratio on fundoscopy (not by OCT reading) greater than or equal to 0.80.
  3. Intraocular pressure (IOP) greater than or equal to 25 by Goldmann tonometry .12
  4. Retinal Detachment or Retinal Break
  5. Acute ocular infection (i.e., Viral conjunctivitis, corneal ulcer, endophthalmitis)
  6. Optic Atrophy with visual field defect reproducible on confrontation visual field testing..
  7. Exam consistent with Herpes Simplex Virus eye infection
  8. Homonymous hemianopsia, quadrantanopsia, bitemporal hemianopsia, or central scotoma related to cerebral vascular disease by Automated Visual Field testing and confrontation visual field testing.
  9. Acute Angle Closure Glaucoma
  10. Gonioscopy grade 0 (slit) limiting ability to safely dilate patient
  11. Severe Tremor, blepharospasm, or other voluntary or involuntary motor condition that prevents ability to examine patient with slit lamp, OCT, gonioscopy, IOP measurement, fundus photography, and Frequency doubling technology perimetry.
  12. Cognitive impairment sufficient to prevent ability to understand and perform Visual Acuity Test with Tumbling E chart, confrontation visual field, slit lamp exam, or any other ocular exam component.
  13. Optic nerve edema
  14. Active retinopathy or retinitis not attributable to onchocercal disease
  15. History of uveitis not associated with onchocercal disease
  16. Any pre-existing chorioretinal scar or retinal degeneration and other significant retinal pathologies (foveomacular schisis, dystrophies, arterial macroaneurysms etc) involving the macula.
  17. Severe ocular pain, that patient rates as 9 or 10 out of 10 pain.
  18. Best corrected or pinhole visual acuity worse than 6/60 (20/200)
  19. Age related macular degeneration (AMD)
* Significant comorbidities such as renal insufficiency, liver failure, or any other acute or chronic illness identified by study clinicians and investigators that interferes with the participant's ability to go to school or work or perform routine household chores.
* Prior allergic / hypersensitivity reactions or intolerance to IVM, ALB, or DEC.
* Treatment with IVM outside of the study after the pre-treatment clearing dose provided in the Part I study.
* >5 motile Mf in the anterior chamber in either eye at the time of enrollment (after pre-treatment with IVM).
* Any Mf identified in the posterior segment of the eye at the time of enrollment (six months after pre-treatment with IVM).
* Any other condition identified by study clinicians or investigators that may preclude participation in the study.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Weil, MD, Principal Investigator — Washington University School of Medicine; Christopher King, MD, PhD, Principal Investigator — Case Western Reserve University; Nicholas Opoku, MB, CHB, MSC, Principal Investigator — University of Health and Allied Sciences, Hohoe, Ghana
Locations (1):
- University of Health and Allied Sciences, Hohoe, Ghana

IPD SHARING:
Plan to Share IPD: Yes
Datasets used for published results will be shared publicly through a journal or other open source data repository so that the broader scientific community can access it. Only de-identified data will be shared publicly.

REFERENCES:
- [Background] Herricks JR, Hotez PJ, Wanga V, Coffeng LE, Haagsma JA, Basanez MG, Buckle G, Budke CM, Carabin H, Fevre EM, Furst T, Halasa YA, King CH, Murdoch ME, Ramaiah KD, Shepard DS, Stolk WA, Undurraga EA, Stanaway JD, Naghavi M, Murray CJL. The global burden of disease study 2013: What does it mean for the NTDs? PLoS Negl Trop Dis. 2017 Aug 3;11(8):e0005424. doi: 10.1371/journal.pntd.0005424. eCollection 2017 Aug. No abstract available. PMID 28771480
- [Background] Taylor MJ, Awadzi K, Basanez MG, Biritwum N, Boakye D, Boatin B, Bockarie M, Churcher TS, Debrah A, Edwards G, Hoerauf A, Mand S, Matthews G, Osei-Atweneboana M, Prichard RK, Wanji S, Adjei O. Onchocerciasis Control: Vision for the Future from a Ghanian perspective. Parasit Vectors. 2009 Jan 21;2(1):7. doi: 10.1186/1756-3305-2-7. PMID 19154624
- [Background] Zimmerman PA, Dadzie KY, De Sole G, Remme J, Alley ES, Unnasch TR. Onchocerca volvulus DNA probe classification correlates with epidemiologic patterns of blindness. J Infect Dis. 1992 May;165(5):964-8. doi: 10.1093/infdis/165.5.964. PMID 1569351
- [Background] Fischer P, Kipp W, Bamuhiga J, Binta-Kahwa J, Kiefer A, Buttner DW. Parasitological and clinical characterization of Simulium neavei-transmitted onchocerciasis in western Uganda. Trop Med Parasitol. 1993 Dec;44(4):311-21. PMID 8134773
- [Background] Dadzie KY, Bird AC, Awadzi K, Schulz-Key H, Gilles HM, Aziz MA. Ocular findings in a double-blind study of ivermectin versus diethylcarbamazine versus placebo in the treatment of onchocerciasis. Br J Ophthalmol. 1987 Feb;71(2):78-85. doi: 10.1136/bjo.71.2.78. PMID 3548811
- [Background] Semba RD, Donnelly JJ, Young E, Green WR, Scott AL, Taylor HR. Experimental ocular onchocerciasis in cynomolgus monkeys. IV. Chorioretinitis elicited by Onchocerca volvulus microfilariae. Invest Ophthalmol Vis Sci. 1991 Apr;32(5):1499-507. PMID 2016131
- [Background] Taylor HR. Onchocerciasis. Int Ophthalmol. 1990 May;14(3):189-94. doi: 10.1007/BF00158317. PMID 2188920
- [Background] Bird AC, el-Sheikh H, Anderson J, Fuglsang H. Changes in visual function and in the posterior segment of the eye during treatment of onchocerciasis with diethylcarbamazine citrate. Br J Ophthalmol. 1980 Mar;64(3):191-200. doi: 10.1136/bjo.64.3.191. PMID 7387952
- [Background] Duke BO. Human onchocerciasis--an overview of the disease. Acta Leiden. 1990;59(1-2):9-24. PMID 2198761
- [Background] Braun G, McKechnie NM, Connor V, Gilbert CE, Engelbrecht F, Whitworth JA, Taylor DW. Immunological crossreactivity between a cloned antigen of Onchocerca volvulus and a component of the retinal pigment epithelium. J Exp Med. 1991 Jul 1;174(1):169-77. doi: 10.1084/jem.174.1.169. PMID 2056276
- [Background] Chandrashekar R, Curtis KC, Weil GJ. Molecular characterization of a parasite antigen in sera from onchocerciasis patients that is immunologically cross-reactive with human keratin. J Infect Dis. 1995 Jun;171(6):1586-92. doi: 10.1093/infdis/171.6.1586. PMID 7539474
- [Background] Chandrashekar R, Ogunrinade AF, Alvarez RM, Kale OO, Weil GJ. Circulating immune complex-associated parasite antigens in human onchocerciasis. J Infect Dis. 1990 Nov;162(5):1159-64. doi: 10.1093/infdis/162.5.1159. PMID 2230240
- [Background] Greene BM, Gbakima AA, Albiez EJ, Taylor HR. Humoral and cellular immune responses to Onchocerca volvulus infection in humans. Rev Infect Dis. 1985 Nov-Dec;7(6):789-95. doi: 10.1093/clinids/7.6.789. PMID 4070916
- [Background] Johnson TP, Tyagi R, Lee PR, Lee MH, Johnson KR, Kowalak J, Elkahloun A, Medynets M, Hategan A, Kubofcik J, Sejvar J, Ratto J, Bunga S, Makumbi I, Aceng JR, Nutman TB, Dowell SF, Nath A. Nodding syndrome may be an autoimmune reaction to the parasitic worm Onchocerca volvulus. Sci Transl Med. 2017 Feb 15;9(377):eaaf6953. doi: 10.1126/scitranslmed.aaf6953. PMID 28202777
- [Background] Kawabata M, Izui S, Anan S, Kondo S, Fukumoto S, Flores GZ, Kobayakawa T. Circulating immune complexes and their possible relevance to other immunological parameters in Guatemalan onchocerciasis. Int Arch Allergy Appl Immunol. 1983;72(2):128-33. doi: 10.1159/000234854. PMID 6874107
- [Background] Semba RD, Murphy RP, Newland HS, Awadzi K, Greene BM, Taylor HR. Longitudinal study of lesions of the posterior segment in onchocerciasis. Ophthalmology. 1990 Oct;97(10):1334-41. doi: 10.1016/s0161-6420(90)32413-2. PMID 2243684
- [Background] Banla M, Tchalim S, Karabou PK, Gantin RG, Agba AI, Kere-Banla A, Helling-Giese G, Heuschkel C, Schulz-Key H, Soboslay PT. Sustainable control of onchocerciasis: ocular pathology in onchocerciasis patients treated annually with ivermectin for 23 years: a cohort study. PLoS One. 2014 Jun 2;9(6):e98411. doi: 10.1371/journal.pone.0098411. eCollection 2014. PMID 24887413
- [Background] Rodriguez-Perez MA, Fernandez-Santos NA, Orozco-Algarra ME, Rodriguez-Atanacio JA, Dominguez-Vazquez A, Rodriguez-Morales KB, Real-Najarro O, Prado-Velasco FG, Cupp EW, Richards FO Jr, Hassan HK, Gonzalez-Roldan JF, Kuri-Morales PA, Unnasch TR. Elimination of Onchocerciasis from Mexico. PLoS Negl Trop Dis. 2015 Jul 10;9(7):e0003922. doi: 10.1371/journal.pntd.0003922. eCollection 2015. PMID 26161558
- [Background] Diawara L, Traore MO, Badji A, Bissan Y, Doumbia K, Goita SF, Konate L, Mounkoro K, Sarr MD, Seck AF, Toe L, Touree S, Remme JH. Feasibility of onchocerciasis elimination with ivermectin treatment in endemic foci in Africa: first evidence from studies in Mali and Senegal. PLoS Negl Trop Dis. 2009 Jul 21;3(7):e497. doi: 10.1371/journal.pntd.0000497. PMID 19621091
- [Background] Zarroug IM, Hashim K, ElMubark WA, Shumo ZA, Salih KA, ElNojomi NA, Awad HA, Aziz N, Katabarwa M, Hassan HK, Unnasch TR, Mackenzie CD, Richards F, Higazi TB. The First Confirmed Elimination of an Onchocerciasis Focus in Africa: Abu Hamed, Sudan. Am J Trop Med Hyg. 2016 Nov 2;95(5):1037-1040. doi: 10.4269/ajtmh.16-0274. Epub 2016 Jun 27. PMID 27352878
- [Background] Eisenbarth A, Achukwi MD, Renz A. Ongoing Transmission of Onchocerca volvulus after 25 Years of Annual Ivermectin Mass Treatments in the Vina du Nord River Valley, in North Cameroon. PLoS Negl Trop Dis. 2016 Feb 29;10(2):e0004392. doi: 10.1371/journal.pntd.0004392. eCollection 2016 Feb. PMID 26926855
- [Background] Katabarwa MN, Eyamba A, Nwane P, Enyong P, Kamgno J, Kuete T, Yaya S, Aboutou R, Mukenge L, Kafando C, Siaka C, Mkpouwoueiko S, Ngangue D, Biholong BD, Andze GO. Fifteen years of annual mass treatment of onchocerciasis with ivermectin have not interrupted transmission in the west region of cameroon. J Parasitol Res. 2013;2013:420928. doi: 10.1155/2013/420928. Epub 2013 Apr 17. PMID 23691275
- [Background] Evans DS, Unnasch TR, Richards FO. Onchocerciasis and lymphatic filariasis elimination in Africa: it's about time. Lancet. 2015 May 30;385(9983):2151-2. doi: 10.1016/S0140-6736(15)61022-4. No abstract available. PMID 26068266
- [Background] Fischer PU, King CL, Jacobson JA, Weil GJ. Potential Value of Triple Drug Therapy with Ivermectin, Diethylcarbamazine, and Albendazole (IDA) to Accelerate Elimination of Lymphatic Filariasis and Onchocerciasis in Africa. PLoS Negl Trop Dis. 2017 Jan 5;11(1):e0005163. doi: 10.1371/journal.pntd.0005163. eCollection 2017 Jan. No abstract available. PMID 28056015
- [Background] Taylor HR, George T. Microfilaria in the cornea in onchocerciasis. Trans R Soc Trop Med Hyg. 1987;81(1):148. doi: 10.1016/0035-9203(87)90308-7. No abstract available. PMID 3445302
- [Background] Greene BM, Taylor HR, Brown EJ, Humphrey RL, Lawley TJ. Ocular and systemic complications of diethylcarbamazine therapy for onchocerciasis: association with circulating immune complexes. J Infect Dis. 1983 May;147(5):890-7. doi: 10.1093/infdis/147.5.890. PMID 6842023
- [Background] Greene BM, Taylor HR, Cupp EW, Murphy RP, White AT, Aziz MA, Schulz-Key H, D'Anna SA, Newland HS, Goldschmidt LP, et al. Comparison of ivermectin and diethylcarbamazine in the treatment of onchocerciasis. N Engl J Med. 1985 Jul 18;313(3):133-8. doi: 10.1056/NEJM198507183130301. PMID 3892293
- [Background] Basanez MG, Pion SD, Boakes E, Filipe JA, Churcher TS, Boussinesq M. Effect of single-dose ivermectin on Onchocerca volvulus: a systematic review and meta-analysis. Lancet Infect Dis. 2008 May;8(5):310-22. doi: 10.1016/S1473-3099(08)70099-9. PMID 18471776
- [Background] Taylor HR, Murphy RP, Newland HS, White AT, D'Anna SA, Keyvan-Larijani E, Aziz MA, Cupp EW, Greene BM. Treatment of onchocerciasis. The ocular effects of ivermectin and diethylcarbamazine. Arch Ophthalmol. 1986 Jun;104(6):863-70. doi: 10.1001/archopht.1986.01050180097039. PMID 3521559
- [Background] Awadzi K, Opoku NO, Attah SK, Lazdins-Helds J, Kuesel AC. A randomized, single-ascending-dose, ivermectin-controlled, double-blind study of moxidectin in Onchocerca volvulus infection. PLoS Negl Trop Dis. 2014 Jun 26;8(6):e2953. doi: 10.1371/journal.pntd.0002953. eCollection 2014 Jun. PMID 24968000
- [Background] Taylor HR. Ivermectin treatment of ocular onchocerciasis. Acta Leiden. 1990;59(1-2):201-6. PMID 2198751
- [Background] Taylor HR, Semba RD, Newland HS, Keyvan-Larijani E, White A, Dukuly Z, Greene BM. Ivermectin treatment of patients with severe ocular onchocerciasis. Am J Trop Med Hyg. 1989 May;40(5):494-500. doi: 10.4269/ajtmh.1989.40.494. PMID 2658637
- [Background] Thomsen EK, Sanuku N, Baea M, Satofan S, Maki E, Lombore B, Schmidt MS, Siba PM, Weil GJ, Kazura JW, Fleckenstein LL, King CL. Efficacy, Safety, and Pharmacokinetics of Coadministered Diethylcarbamazine, Albendazole, and Ivermectin for Treatment of Bancroftian Filariasis. Clin Infect Dis. 2016 Feb 1;62(3):334-341. doi: 10.1093/cid/civ882. Epub 2015 Oct 20. PMID 26486704
- [Background] Awadzi K, Gilles HM. Diethylcarbamazine in the treatment of patients with onchocerciasis. Br J Clin Pharmacol. 1992 Oct;34(4):281-8. doi: 10.1111/j.1365-2125.1992.tb05632.x. No abstract available. PMID 1457260
- [Background] Opoku NO, Bakajika DK, Kanza EM, Howard H, Mambandu GL, Nyathirombo A, Nigo MM, Kasonia K, Masembe SL, Mumbere M, Kataliko K, Larbelee JP, Kpawor M, Bolay KM, Bolay F, Asare S, Attah SK, Olipoh G, Vaillant M, Halleux CM, Kuesel AC. Single dose moxidectin versus ivermectin for Onchocerca volvulus infection in Ghana, Liberia, and the Democratic Republic of the Congo: a randomised, controlled, double-blind phase 3 trial. Lancet. 2018 Oct 6;392(10154):1207-1216. doi: 10.1016/S0140-6736(17)32844-1. Epub 2018 Jan 18. PMID 29361335
- [Background] Bird AC, Anderson J, Fuglsang H. Morphology of posterior segment lesions of the eye in patients with onchocerciasis. Br J Ophthalmol. 1976 Jan;60(1):2-20. doi: 10.1136/bjo.60.1.2. PMID 1268156
- [Background] Fuglsang H, Anderson J. Further observations on the relationship between ocular onchocerciasis and the head nodule, and on the possible benefit of nodulectomy. Br J Ophthalmol. 1978 Jul;62(7):445-9. doi: 10.1136/bjo.62.7.445. PMID 678496
- [Background] Wojtkowski M, Bajraszewski T, Gorczynska I, Targowski P, Kowalczyk A, Wasilewski W, Radzewicz C. Ophthalmic imaging by spectral optical coherence tomography. Am J Ophthalmol. 2004 Sep;138(3):412-9. doi: 10.1016/j.ajo.2004.04.049. PMID 15364223
- [Background] Jolodar A, Fischer P, Buttner DW, Miller DJ, Schmetz C, Brattig NW. Onchocerca volvulus: expression and immunolocalization of a nematode cathepsin D-like lysosomal aspartic protease. Exp Parasitol. 2004 Jul-Aug;107(3-4):145-56. doi: 10.1016/j.exppara.2004.06.006. PMID 15363940
- [Background] Donner A, Koval JJ. A multivariate analysis of family data. Am J Epidemiol. 1981 Jul;114(1):149-54. doi: 10.1093/oxfordjournals.aje.a113162. PMID 7246523
- [Background] Rutterford C, Copas A, Eldridge S. Methods for sample size determination in cluster randomized trials. Int J Epidemiol. 2015 Jun;44(3):1051-67. doi: 10.1093/ije/dyv113. Epub 2015 Jul 13. PMID 26174515
- [Derived] Opoku NO, Doe F, Dubben B, Fetcho N, Fischer K, Fischer PU, Gordor S, Goss CW, Gyasi ME, Hoerauf A, Hong AR, Kanza E, King CL, Laryea R, Lew D, Seidu MA, Weil GJ. A randomized, open-label study of the tolerability and efficacy of one or three daily doses of ivermectin plus diethylcarbamazine and albendazole (IDA) versus one dose of ivermectin plus albendazole (IA) for treatment of onchocerciasis. PLoS Negl Trop Dis. 2023 May 19;17(5):e0011365. doi: 10.1371/journal.pntd.0011365. eCollection 2023 May. PMID 37205721

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited in the Nkwanta North District in the Volta Region in Ghana through open community meetings.
Period: Baseline
Arm/Group | IVM + ALB | IDA x 1 Dose | IDA x 3 Doses
Started | 52 | 51 | 51
Completed | 52 | 51 | 51
Not Completed | 0 | 0 | 0
Period: Month 3
Arm/Group | IVM + ALB | IDA x 1 Dose | IDA x 3 Doses
Started | 52 | 51 | 51
Completed | 52 | 51 (1 participant was not able to be followed up with at Month 3, but was seen at Month 12 and 18) | 50
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Period: Month 12
Arm/Group | IVM + ALB | IDA x 1 Dose | IDA x 3 Doses
Started | 52 | 51 | 50
Completed | 51 | 50 | 48
Not Completed | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Death | 1 | 1 | 0
Period: Month 18
Arm/Group | IVM + ALB | IDA x 1 Dose | IDA x 3 Doses
Started | 51 | 50 | 48
Completed | 45 | 50 (Previous participant who was loss to follow up was able to complete the 18 month time point) | 48
Not Completed | 6 | 0 | 0
Not completed — Lost to Follow-up | 6 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVM + ALB | IDA x 1 Dose | IDA x 3 Doses | Total
Number analyzed (Participants) | 52 | 51 | 51 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (12.18) | 38.52 (14.08) | 37.65 (2.16) | 37.65 (13.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 11 | 50
  Male | 31 | 33 | 40 | 104
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Ghana | 52 | 51 | 51 | 154
Ocular Microfilarae positive [Count of Participants; unit: Participants] — Presence of microfilariae in the anterior or posterior chamber of the eye at baseline
  Participants
    Positive for ocular microfilarae | 2 | 2 | 0 | 4
    Negative for ocular microfilarae | 50 | 49 | 51 | 150

OUTCOME MEASURES:

1. Primary Outcome: Rates of Severe Adverse Events (SAEs) Across Study Arms
Description: Rates of severe adverse events (grade 3 or higher) following 1-day or 3-day triple drug treatment will be compared against those of the comparator regimen of 1 day of IVM/ALB.
Time Frame: Within 7 days following end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | IVM + ALB | IDA x 1 Dose | IDA x 3 Doses
Number analyzed (Participants) | 52 | 51 | 51
Participants | 0 | 0 | 0

2. Primary Outcome: Percentage of Worms Killed Across Study Arms
Description: The effect of three treatment regimens for killing adult female O. volvulus worms will be compared based on the percentage of all adult female worms in nodules that are alive with embryos in the uterus 18 months after treatment.
Time Frame: 18 months following treatment.
Population: The analysis was conducted on worms from participants who had nodulectomies conducted at 18 months. Not all participants who completed the study had nodulectomies conducted.
Measure: Count of Units; unit: Female worms in nodules
Units Other Than Participants: Female worms in nodules
Arm/Group | IVM + ALB | IDA x 1 Dose | IDA x 3 Doses
Number analyzed (Participants) | 41 | 46 | 47
Number analyzed (Female worms in nodules) | 196 | 274 | 300
Female worms in nodules | 127 | 142 | 159
Statistical Analysis 1: Comparison: IVM + ALB vs IDA x 1 Dose; IA vs IDA for living female O. volvulus worms in nodules after treatment; Test type: Superiority; p = 0.192, Regression, Logistic — Participant level random effects were included in the model to adjust for multiple worms/person. Adjusted P values were model-adjusted for repeated measurements per person; Mixed-effects logistic regression model where study participant was included as a random effect to adjust for multiple worms per person; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.84 to 2.38]
Statistical Analysis 2: Comparison: IVM + ALB vs IDA x 3 Doses; IA vs IDA3 for living female O. volvulus worms in nodules after treatment; Test type: Superiority; p = 0.107, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.92 to 2.29]
Statistical Analysis 3: Comparison: IVM + ALB vs IDA x 1 Dose vs IDA x 3 Doses; Test type: Superiority — IA vs IDA treatment groups for living female O. volvulus worms in nodules after treatment; p = 0.068, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.97 to 2.15]
Statistical Analysis 4: Comparison: IDA x 1 Dose vs IDA x 3 Doses; IDA vs IDA3 for living female O. volvulus worms in nodules after treatment; Test type: Superiority; p = 0.918, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.59 to 1.79]

3. Secondary Outcome: Rates of SAEs by Treatment Group in Those With Intraocular Microfilariae Just Prior to Treatment With IDA
Description: Rates of adverse events grade 3 or higher that occur within 7 days of treatment in the subset of participants who have intraocular microfilariae just prior to treatment with IDA will be compared by treatment group.
Time Frame: within 7 days following end of treatment
Population: For the Arm IDA x 3 doses, no participants had intraocular microfilariae present at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | IVM + ALB | IDA x 1 Dose | IDA x 3 Doses
Number analyzed (Participants) | 2 | 2 | 0
Participants | 0 | 0 | 0

4. Secondary Outcome: Rates of Ocular Adverse Events (Any Grade) by Treatment Group
Description: Rates of ocular adverse events of any grade within 3 months will be compared by treatment group.
Time Frame: within 3 months of treatment with IDA
Measure: Count of Participants; unit: Participants
Arm/Group | IVM + ALB | IDA x 1 Dose | IDA x 3 Doses
Number analyzed (Participants) | 52 | 51 | 51
Participants | 4 | 4 | 3

5. Secondary Outcome: Effectiveness of Killing Adult Female Worms
Description: The effectiveness of three treatment regimens for killing adult female O. volvulus worms based on the percentage of all adult female worms in nodules that are alive 18 months after treatment.
Time Frame: 18 months following treatment
Population: Analysis conducted on participants who had nodulectomies conducted at 18 months. Not all participants who completed the study had nodulectomies conducted.
Measure: Count of Units; unit: Female worms in nodule
Units Other Than Participants: Female worms in nodule
Arm/Group | IVM + ALB | IDA x 1 Dose | IDA x 3 Doses
Number analyzed (Participants) | 41 | 46 | 47
Number analyzed (Female worms in nodule) | 198 | 274 | 300
Female worms in nodule | 127 | 142 | 159
Statistical Analysis 1: Comparison: IVM + ALB vs IDA x 1 Dose; IA vs IDA for living female O. volvulus worms in nodules after treatment; Test type: Superiority; p = 0.192, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.84 to 2.38]
Statistical Analysis 2: Comparison: IVM + ALB vs IDA x 3 Doses; IA vs IDA3 for living female O. volvulus worms in nodules after treatment; Test type: Superiority; p = 0.107, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.92 to 2.29]
Statistical Analysis 3: Comparison: IVM + ALB vs IDA x 1 Dose vs IDA x 3 Doses; IA vs IDA groups for living female O. volvulus worms in nodules after treatment; Test type: Superiority; p = 0.068, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.97 to 2.15]
Statistical Analysis 4: Comparison: IDA x 1 Dose vs IDA x 3 Doses; IDA vs IDA3 for living female O. volvulus worms in nodules after treatment; Test type: Superiority; p = 0.918, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.59 to 1.79]

6. Secondary Outcome: Effectiveness of Clearing Microfilariae From Skin by Skin Snips
Description: The effectiveness of three treatment regimens for complete clearance of microfilariae from the skin as determined by skin snips at 3, 12, and 18 months after treatment with IDA will be compared by treatment arm.
Time Frame: Baseline, 3 months, 12 months, & 18 months following treatment.
Measure: Geometric Mean (95% Confidence Interval); unit: Count of Skin Microfilaria
Arm/Group | IVM + ALB | IDA x 1 Dose | IDA x 3 Doses
Number analyzed (Participants) | 52 | 51 | 51
Count of Skin Microfilaria
  Baseline | 3.1 [1.8 to 5.5] | 1.7 [0.8 to 3.6] | NA [NA to NA] — Geometric mean could not be estimated because all values were zero
  Month 3 | 1.9 [1.0 to 3.4] | 3 [NA to NA] — 95% CI could not be estimated because raw data had only one nonzero value | 2.1 [0.9 to 4.7]
  Month 12 | 4.9 [2.8 to 8.5] | 2.5 [1.6 to 3.8] | 4.7 [2.8 to 7.9]
  Month 18 | 7.0 [3.6 to 13.9] | 9.0 [4.6 to 17.6] | 8.6 [4.3 to 17.1]

7. Secondary Outcome: Effectiveness for Preventing Reappearance of Microfilariae in the Skin by Skin Snips
Description: The effectiveness of three treatment regimens for preventing reappearance of microfilariae in the skin as determined by skin snips at 12 and 18 months after treatment will be compared by treatment arm. Measured by the presence of microfilariae in skin snips.
Time Frame: Baseline, 12 months, and 18 months following treatment
Measure: Number; unit: Count of microfilarae+ participants
Arm/Group | IVM + ALB | IDA x 1 Dose | IDA x 3 Doses
Number analyzed (Participants) | 52 | 51 | 51
Count of microfilarae+ participants
  Baseline | 7 | 6 | 0
  Month 12 | 23 | 21 | 21
  Month 18 | 20 | 15 | 17

8. Primary Outcome: Percentage of Worms Sterilized Across Study Arms
Description: The effect of three treatment regimens for sterilizing adult female O. volvulus worms will be compared based on the percentage of all adult female worms that are fertile in the nodules 18 months after treatment.
Time Frame: 18 months following treatment.
Population: The analysis was conducted on worms from participants who had nodulectomies conducted at 18 months. Not all participants who completed the study had nodulectomies conducted. Female worms were excluded who had collapsed uteri that could not be evaluated for fertility.
Measure: Count of Units; unit: Female worms with intact uterus
Units Other Than Participants: Female worms with intact uterus
Arm/Group | IVM + ALB | IDA x 1 Dose | IDA x 3 Doses
Number analyzed (Participants) | 41 | 46 | 47
Number analyzed (Female worms with intact uterus) | 180 | 261 | 281
Female worms with intact uterus | 41 | 40 | 34
Statistical Analysis 1: Comparison: IVM + ALB vs IDA x 1 Dose; IA vs IDA in fertile female O. volvulus worms in nodules after treatment; Test type: Superiority; p = 0.134, Regression, Logistic — Adjusted p values were model-adjusted for repeated measurements per person. Participant level random effects were included in the model to adjust for multiple worms/person; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.85 to 3.21]
Statistical Analysis 2: Comparison: IVM + ALB vs IDA x 3 Doses; IA vs IDA3 for fertile female O. volvulus worms in nodules after treatment; Test type: Superiority; p = 0.023, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.23, 95% CI 2-sided [1.12 to 4.44]
Statistical Analysis 3: Comparison: IDA x 1 Dose vs IDA x 3 Doses; IDA1 vs IDA3 for fertile female O. volvulus worms in nodules after treatment; Test type: Superiority; p = 0.430, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.32, 95% CI 2-sided [.64 to 2.85]
Statistical Analysis 4: Comparison: IVM + ALB vs IDA x 1 Dose vs IDA x 3 Doses; IA vs IDA treatment groups for fertile female O. volvulus worms in nodules after treatment; Test type: Superiority; p = 0.023, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.91, 95% CI 2-sided [1.09 to 3.34]

ADVERSE EVENTS:
Time Frame: Data was collected on adverse events for safety from baseline to 3 months after treatment. Serious adverse events and mortality were collected throughout the trial from baseline to 18 months after treatment.
Arm/Group | IVM + ALB | IDA x 1 Dose | IDA x 3 Doses
All-Cause Mortality (participants affected / at risk) | 1/52 | 1/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 11/52 | 15/51 | 11/51
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVM + ALB (N=52) | IDA x 1 Dose (N=51) | IDA x 3 Doses (N=51)
Chills (General disorders) | 1 (1) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Itching skin (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 4 (4)
Joint or muscle pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2)
Itching, ocular (Eye disorders) | 4 (4) | 1 (1) | 2 (2)
Waist Pain (General disorders) | 2 (2) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
Pause on clinical trial operations between March 2020 - June 2020 due to the COVID-19 pandemic. Decreased health and viability of the adult female worm population in participants may have reduced the study's ability to detect a significant macrofilaricidal effect of IDA. Study enrolled participants with light/moderate infections, which greatly decreased the risk of SAEs occurring. Future studies to assess tolerability of IDA would need to be conducted with higher infection rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT04188301/Prot_SAP_001.pdf